| <b>RECOVER Web Por</b> | ta |
|------------------------|----|
| Template Content | ٧Ź |

Implementation of a Clinical Pathway for Paediatric Concussion in Acute Care Settings:
Measuring Health Outcomes of the RECOVER Intervention Project

REB18-0405

21.June.2018

## Home page:

Welcome to the **RECOVER** site! RECOVER offers information and resources on concussion in children to help families better understand common symptoms associated with concussion, where and when to seek medical care, and how to self-monitor or manage symptoms to promote optimal recovery. The

RECOVER site also offers a tool to allow youth with concussion, as well as caregivers, to **track recovery** by reporting and monitoring symptom ratings.

Click here to learn more!

## About page:

#### THE RECOVER STUDY

RECOVER (Resources on Concussion in a Virtual Environment) is a study conducted by researchers at the University of Calgary and University of Alberta. To improve and standardize care for children with concussion who are seen in emergency departments, this study has developed tools to help clinicians and families to learn more about, assess, and monitor concussion. Key tools include a clinical pathway to guide clinicians in providing concussion care and a web portal for families that provides up-to-date and reliable information on concussion. The RECOVER study will evaluate the effects of introducing these new elements into routine concussion care for children in emergency departments. The ultimate goal of the study is to improve the health outcomes of youth diagnosed with concussion by providing up-to-date and reliable evidence-based information on concussion symptoms, management, and follow-up care.

## **REGISTER TO PARTICIPATE!**

Looking for a tool to help you (or your child) **track your recovery?** The RECOVER site can help you identify common concussion symptoms and to monitor your own symptoms in order to promote optimal recovery. We are currently looking for youth and caregivers to enroll in the RECOVER study. If you (or your child) have recently been diagnosed with concussion in an emergency department at one of the following clinical sites:

- Alberta Children's Hospital (Calgary)
- South Health Campus (Calgary)
- Stollery Children's Hospital (Edmonton)
- North East Community Health Centre (Edmonton)
- Grey Nuns' Community Hospital (Edmonton)

**SIGN UP NOW!** 

Please read the options below carefully and select one to create an account.

**OPTION 1: Participate Linkage** 

Click here for study enrolment options

with Consent for Data

In order to better understand the short- and long-term health outcomes of children with concussion, the RECOVER study would like to link information that you provide on this web portal about your concussion symptoms and recovery with your personal health information collected by Alberta Health Services. Health information collected for this study will be limited to health utilization data (e.g., visits to clinics, use of diagnostic services) and basic sociodemographic information (e.g., geography, age, gender). All personal health information will be kept strictly confidential and be used only for the purpose of this study. >> Click here for more information on the study and authorization to use your health information.

# **OPTION 2: Participate Anonymously**

You may also wish to participate in the study but remain anonymous. This means that the responses you provide on the web portal will not be linked to your personal health information collected by Alberta Health Services. You will still receive all information available on the RECOVER site that is pertinent to concussion to help you track your recovery. Keep in mind, however, that this option will give us less of a clear picture on health outcomes associated with the information provided on this site.

| To enroll in the study, please choose one of the following: |
|---|
| ☐ I wish to enroll in the RECOVER study and authorize use of my health information collected by Alberta Health Services |
| ☐ I wish to enroll in the RECOVER study and remain anonymous (I do not authorize use of my health information collected by Alberta Health Services) |
| ☐ I have read and accept the consent form that describes the purpose of the study and the conditions for authorizing use of my health information |
| PREVIOUS RESEARCH PARTCIPATION: |
| Have you participated in any other research studies on concussion? |
| ☐ Yes ☐ No If yes, please specify name of study: |
| Click here to create an account |

#### FOR MORE INFORMATION

Study Coordinator: Anh Ly Email: recover@ucalgary.ca Phone number: 403-955-5442

| Consent Form: | |
|---|---|
| Approval Date: | _ |
| Expiration Date: | <u>-</u> |
| REB Study ID: | _ |
| Protocol Title: RECOVER Pediatr | ic Concussion Clinical Pathway Intervention Project |
| Principal Investigator: Dr. Keith | Yeates, Department of Psychology, University of Calgary |
| Sponsors: 1) Alberta Health Serv | vices; 2) Brain Canada |

**DESCRIPTION**: You are invited to participate in a research study on the implementation of a clinical pathway to standardize concussion care for children seen in emergency departments. This study is being conducted at five clinical sites in Calgary and Edmonton, Alberta. The purpose of the study is to improve the health outcomes of youth diagnosed with concussion by providing up-to-date and reliable evidencebased information on concussion symptoms, management, and follow-up care. You were selected as a possible participant in this study because you (or your child) have recently visited an emergency department and were diagnosed with concussion by a physician. As part of this study, we will ask you to complete questionnaires about your (or your child's) experience with concussion, such as self-ratings of your symptoms, satisfaction with care in the emergency department, and the impacts of concussion on your daily life. If you have participated in previous studies on concussion through the University of Calgary or University of Alberta that were led by Dr. Keith Yeates, we will ask for permission to access important data collected about your (or your child's) concussion during his or her previous participation in this research in order to better understand the variables associated with recovery from concussion. We would also like to link information that you provide on the RECOVER web portal with your personal health information collected by Alberta Health Services in order to better understand health utilization patterns as well as health outcomes of children with concussion. You may, however, opt to participate anonymously in the study, which means that your responses on the web portal will not be linked to your personal health information collected by Alberta Health Services.

**TIME INVOLVEMENT**: Your participation will vary depending on the course of your recovery and improvements in symptoms. The questionnaires that you will be asked to complete will take approximately 5-10 minutes each to complete. Three questionnaires will be administered only once, and one questionnaire will be administered on a weekly basis (with option to complete daily) until you report full recovery.

RISKS AND BENEFITS: The risks associated with this study are minimal and include some fatigue and/or psychological discomfort from completion of the questionnaires. There are no direct benefits to you (or your child) for participating in this project, nor are there any costs or payments involved in order to participate. An indirect benefit of this study is that you may find the symptom/recovery tracking tool that we developed to be helpful to give you some information on the trajectory of your symptom ratings in comparison to average recovery rates for children of the same age.

**PAYMENTS**: You will not receive any payment for your participation.

**PARTICIPANT'S RIGHTS**: If you have read this form and have decided to participate in this study, please understand that your participation is voluntary and you have the right to withdraw your consent or

discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled. You also have the right to refuse to answer particular questions. Your individual privacy will be maintained in all published and written data resulting from this study.

**AUTHORIZATION TO USE YOUR HEALTH INFORMATION FOR RESEARCH PURPOSES**: Because information about you and your health is personal and private, it generally cannot be used in this research study without your authorization. The form is intended to inform you about how your health information will be used or disclosed in the study. Your information will only be used in accordance with this authorization form and the informed consent. Please read it carefully before agreeing.

**HOW WILL MY HEALTH INFORMATION BE UTILIZED IN THE STUDY?**: The purpose of this study is to collect information about concussion in children and youth. We are interested in understanding more about recovery rates, satisfaction with care, impacts of concussion on daily activities, health utilization patterns, health care costs, and the impact of an educational intervention tool for families. Your health information may be used in scientific publications. The results of this research study may be presented at scientific or medical meetings. However, your identity will not be disclosed.

WHAT PERSONAL INFORMATION WILL BE OBTAINED, USED, OR DISCLOSED?: Your health information related to this study may be used or disclosed in connection with this research study, including, but not limited to, your electronic email address, year of birth, demographic information, and health services utilization.